CLINICAL TRIAL: NCT00259493
Title: Graft Patency Following Off-Pump CABG Vs. On-Pump CABG Using 64 MDCT Bypass Graft CT Angiography
Brief Title: Graft Patency in Beating Heart Vs. Conventional CABG Using Cardiac CT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Trillium Health Centre (Other)
Collaborators: Toshiba America Medical Systems, Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2005-11-25; First posted 2005-11-29 (Estimated); Last update posted 2006-09-11 (Estimated); Status verified 2005-09

CONDITIONS: Coronary Artery Disease Amenable to Bypass Graft Surgery
Keywords: Coronary Artery Disease; Coronary Artery Bypass Graft Surgery; Off-pump CABG; Cardiac CT; Bypass Graft CT angiography
MeSH Terms: conditions — Coronary Artery Disease

INTERVENTIONS:
Procedure: Off-Pump Coronary Artery Bypass Graft Surgery

SUMMARY:
The purpose of this study is to compare graft patency rates following coronary artery bypass graft surgery performed by beating heart vs. conventional techniques using cardiac CT scanning to evaluate the bypass grafts.

DETAILED DESCRIPTION:
The issue of whether to perform conventional CABG or off-pump CABG continues to be the subject of debate. Controversy remains regarding the appropriateness of applying OPCAB to all patients as opposed to selected sub-populations.

The main strategy of CABG is to obtain complete revascularization with the least morbidity and highest long-term patency rates. Current medical literature is conflicted regarding graft patency rates in OPCAB vs. conventional CABG. Data is also limited due to patient refusal for conventional angiography to assess grafts following surgery. Cardiac computed tomography (CT) offers a non-invasive method to assess graft patency that is 100% accurate for the diagnosis of graft patency vs. occlusion. This study is a prospective randomized controlled trial evaluating graft patency in on-pump vs. off-pump CABG using cardiac CT scanning. The study hypothesis is that graft patency rates will be equivalent between the two techniques.

ELIGIBILITY:
Inclusion Criteria:

* Surgery indicated
* Patient is hemodynamically stable
* Isolated coronary artery surgery (no valve)
* No contraindications to cardiopulmonary bypass
* No previous surgery (not redo CABG)

Exclusion Criteria:

* critically ill patient with hemodynamic instability.
* concomitant cardiac procedures.
* inability to provide written informed consent.
* prior severe reaction to contrast dye :
* life-threatening anaphylactoid reactions
* cardiac dysrhythmias and arrest
* cardiovascular and pulmonary collapse
* elevated serum creatinine (>150 mmol/L).
* contraindications to cardiopulmonary bypass.
* Age < 18 years .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350
Dates: Start 2005-12; Study Completion 2007-10

PRIMARY OUTCOMES:
Graft patency as determined by bypass graft CT angiography at 3 months and 12 months following surgery

SECONDARY OUTCOMES:
Length of Hospital Stay
Blood Loss
Operative Time
Post-op Complications
Quality of Life Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Tarang N Sheth, MD, FRCPC, Principal Investigator — Trillium Health Centre; Gopal Bhatnagar, MD, FRCSC, Principal Investigator — Trillium Health Centre
Locations (1):
- Trillium Health Centre, Mississauga, Ontario, Canada